CLINICAL TRIAL: NCT02661932
Title: Efficiency and Safety Study of Ovarian Stimulation With Letrozole for Fertility Preservation in Breast Cancer Patients
Brief Title: Fertility Preservation in Breast Cancer Patients
Acronym: Brovale
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BC-POF 2012
Record Dates: First submitted 2015-12-23; First posted 2016-01-25 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms; Fertility
Keywords: Fertility preservation; letrozole; Ovarian stimulation
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole associated COS (Experimental): Breast cancer patients undergo fertility preservation with letrozole associated COS for oocyte collection.
  Letrozole is administered orally (5mg/day) during the entire stimulation protocol until ovulation triggering.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Patients start ovarian stimulation protocol according to their menstrual cycle phase at enrollment (standard or "random start"). Ovarian stimulation includes gonadotropins administration in a GnRH antagonist protocol Standard Protocol: letrozole is orally administered 2 tablets per day (2,5mgx2/d) from cycle day 2 throughout the ovarian stimulation with gonadotropins protocol until ovulation triggering. GnRH antagonist is administered as soon as at least one follicle reaches 14 mm.
  "Random start" protocol: letrozole is administered throughout the stimulation together with gonadotropins and GnRH antagonist, until ovulation triggering.
  Oocytes are collected 36h after ovulation triggering. All patients receive GnRH antagonist after oocyte retrieval for 3-7 days or until chemotherapy starts, to induce luteolysis.
  Other Names: Femara

SUMMARY:
The purpose of this study is to evaluate efficiency and safety of controlled ovarian stimulation (COS) associated with an aromatase inhibitor (letrozole) for fertility preservation in breast cancer patients.

DETAILED DESCRIPTION:
Patients enrolled in this study undergo standard or "random start" ovarian stimulation with Gonadotropins using antagonist protocol before the beginning of chemotherapy. Ovulation is triggered in all patients with a GnRH agonist since amendment P2015/091 (Decapeptyl 0,2mg).

At oocyte retrieval, aspirated follicular fluid is separated from the flush medium for hormonal assays, and oocytes are denuded for ICSI(Intra Cytoplasmic Sperm Injection) or vitrification. Cumulus cells are collected for subsequent analysis of oocyte quality gene expression.

A. Primary objective of the study is to evaluate efficiency of letrozole associated ovarian stimulation for fertility preservation in breast cancer patients in terms of oocyte maturation rate.

Patients' results for primary endpoint are prospectively compared to infertile patients undergoing COS without letrozole.

B. Secondary objectives of the study aim to evaluate safety of the protocol:

1. Estradiol and progesterone levels at ovulation triggering, ovulation and during luteal phase after oocyte retrieval (days 3 and 8)
2. The risk of disease relapse will be assessed by long-term follow-up of these patients (up to 5 years) as well as an evaluation of circulating tumoral DNA before and after ovarian stimulation.
3. Finally obstetrical outcomes will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer female patients of less than 41 years old
* Addressed to fertility preservation Unit before starting chemotherapy

Exclusion Criteria:

* Metastatic breast cancer
* Known premature ovarian failure
* Basal FSH > 20 IU(International Unit)
* Surgical contra-indications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Oocyte maturation rate | At oocyte collection (48 hours after last administration of letrozole, following COS protocol).
  Following letrozole associated COS, oocytes are collected and evaluated for maturation rate (%).
  These results are prospectively compared to infertile patients undergoing similar COS (GnRH antagonist protocol) without letrozole.

SECONDARY OUTCOMES:
Hormonal levels | during stimulation at ovulation trigger and oocyte retrieval and during luteal phase (days 3 and 8)
  Estradiol and Progesterone levels are measured on serum samples to confirm the effect of COS associated with letrozole on hormonal levels
Circulating tumoral DNA | At enrollment (before letrozole associated COS) and at oocyte retrieval (48 hours after last administration of letrozole, following COS protocol)
  3 EDTA (Ethylene Diamine Tetra-Acetic Acid) tubes are collected for plasma extraction. 1 EDTA tube is collected for whole blood.
  Circulating tumoral DNA will be assessed on plasma samples according to primary tumoral mutation screening. Whole blood will used as reference.
Comparison of breast cancer recurrence rate in patients who underwent letrozole associated COS with an oncological control group | 2 and 5 years after letrozole associated COS
  Oncological follow-up for relapse risk assessment will be carried out at 2 and 5 years of follow-up by medical chart review. Local, contralateral and/or distant recurrence of the disease will be reported.
  These data will be compared to a control group matched for age and type of disease who were diagnosed with breast cancer during the same period but did not undergo letrozole associated COS for fertility preservation.
Ovarian reserve | At enrollment, 2 and 5 years after letrozole associated COS for fertility preservation
  AMH (anti-mullerian hormone) and FSH (follicle stimulating hormone) are assessed on blood samples to evaluate the gonadotoxicity of chemotherapy.
Obstetrical outcome: malformation rate | Through study completion: data collection at 2 and 5 years after letrozole associated COS
  Malformation will be evaluated in patients who conceive with a previously vitrified oocyte (following letrozole associated COS): malformation assessment during prenatal morphology ultrasound and/or at birth
Neonatal outcomes: gestational age at birth | Through study completion: data collection at 2 and 5 years after letrozole associated COS
  Neonatal outcomes will be evaluated in patients who conceive with a previously vitrified oocyte (following letrozole associated COS): gestational age at birth. Preterm delivery is defined by birth < 37 weeks gestation.
Neonatal outcomes: delivery procedure | Through study completion: data collection at 2 and 5 years after letrozole associated COS
  Neonatal outcomes will be evaluated in patients who conceive with a previously vitrified oocyte (following letrozole associated COS). Delivery procedure is defined as spontaneous, instrumental or cesarean section
Neonatal outcomes: birth weight | Through study completion: data collection at 2 and 5 years after letrozole associated COS
  Neonatal outcomes will be evaluated in patients who conceive with a previously vitrified oocyte (following letrozole associated COS). Birth weight will be reported in grams.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Demeestere, Principal Investigator — Erasme-CUB
Locations (1):
- Erasme-CUB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldrat O, De Cooman M, Mailliez A, Delbaere A, D'Orazio E, Demeestere I, Decanter C. Efficacy and safety of controlled ovarian hyperstimulation with or without letrozole for fertility preservation in breast cancer patients: A multicenter retrospective study. Eur J Cancer. 2022 Oct;174:134-141. doi: 10.1016/j.ejca.2022.07.017. Epub 2022 Aug 20. PMID 35998549
- [Result] Goldrat O, Delbaere A, Demeestere I. Impact of letrozole-associated controlled ovarian hyperstimulation on ART outcomes and endocrinological parameters. Hum Reprod. 2022 Oct 31;37(11):2722-2723. doi: 10.1093/humrep/deac206. No abstract available. PMID 36124889
- [Result] Goldrat O, Gervy C, Englert Y, Delbaere A, Demeestere I. Progesterone levels in letrozole associated controlled ovarian stimulation for fertility preservation in breast cancer patients. Hum Reprod. 2015 Sep;30(9):2184-9. doi: 10.1093/humrep/dev155. Epub 2015 Jun 24. PMID 26109617
- [Derived] Goldrat O, Van Den Steen G, Gonzalez-Merino E, Dechene J, Gervy C, Delbaere A, Devreker F, De Maertelaer V, Demeestere I. Letrozole-associated controlled ovarian hyperstimulation in breast cancer patients versus conventional controlled ovarian hyperstimulation in infertile patients: assessment of oocyte quality related biomarkers. Reprod Biol Endocrinol. 2019 Jan 3;17(1):3. doi: 10.1186/s12958-018-0443-x. PMID 30606204